CLINICAL TRIAL: NCT07316205
Title: Beyond Pink: Assessing Gingival Pigmentation in the Egyptian Population: A Cross-Sectional Study
Brief Title: Gingival Pigmentation Intensity and Distribution Among Egyptians
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzahraa Alghriany, Lecturer, Oral medicine, Periodontology and Oral diagnosis, Faculty of dentistry, Assiut University
Other Study IDs: Gingival pigmentation
Record Dates: First submitted 2025-11-24; First posted 2026-01-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gingiva Disorder
Keywords: gingival pigmentation; egyptians
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Evaluate the gingival pigmentation in the anterior zone using the Oral pigmentation index, Hedin melanin index and de Krom classification
  Interventions: Other: Evaluatation of the gingival pigmentation intensty and distribution

INTERVENTIONS:
Other: Evaluatation of the gingival pigmentation intensty and distribution — After taking history & clinical examination, three examiners will evaluate the gingival pigmentation in the anterior zone using the following indices:
  Clinical evaluation:
  Oral pigmentation index (DOPI) Dummet et al.,1967:
  This index of oral pigmentation is the commonly used index due to its simplicity and ease of use measure hyperpigmentation intensity. The scores are as follows:
  * No clinical pigmentation (pink-colored gingiva)
  * Mild clinical pigmentation (mild light brown color)
  * Moderate clinical pigmentation (medium brown or mixed pink and brown color)
  * Heavy clinical pigmentation (deep brown or bluish black color) Hedin melanin index (Hedin.,1977) for distribution of the pigmentation in the gingiva.
  It is scored as:
  0 = no gingival pigmentation.
  1. = one or two solitary units of interdental papillae are pigmented.
  2. = more than 3 separate units of interdental papillae are pigmented.
  3. = 1 short continuous band of pigmented

SUMMARY:
The aim of the present study is to evaluate the distribution, intensity and extension of gingival hyperpigmentation among a sample of Egyptian population.

DETAILED DESCRIPTION:
After taking history & clinical examination, three examiners will evaluate the gingival pigmentation in the anterior zone using the following indices:

Clinical evaluation:

Oral pigmentation index (DOPI):

This index of oral pigmentation is the commonly used index due to its simplicity and ease of use measure hyperpigmentation intensity. The scores are as follows:

* No clinical pigmentation (pink-colored gingiva)
* Mild clinical pigmentation (mild light brown color)
* Moderate clinical pigmentation (medium brown or mixed pink and brown color)
* Heavy clinical pigmentation (deep brown or bluish black color) Hedin melanin index for distribution of the pigmentation in the gingiva.

It is scored as:

0 = no gingival pigmentation.

1. = one or two solitary units of interdental papillae are pigmented.
2. = more than 3 separate units of interdental papillae are pigmented.
3. = 1 short continuous band of pigmented gingiva.
4. = one wideband continuous pigmented gingiva between the canines. The total scores of Hedin index of the mandible and maxilla will be obtained at baseline, one month, and six months after the depigmentation procedures.

de Krom classification:

The de Krom classification will be conceived to assess pigmentation distribution. It includes six categories:

Category 1: Broad zone of pigmentation completely surrounds the dentition, displaying a clear apical contour. Apical to the mucogingival junction, the mucosa is pink. Gingival color can vary from dark to light brown. The zone is symmetric and the color uniform.

Category 2: Narrow zone of non-pigmented gingiva completely surrounds the teeth, that is, the marginal gingiva is pink. The remaining attached gingiva is as in Category 1, a broad zone of pig mentation. The zone is symmetric and the color uniform.

Category 3: Mucosa is completely pink, except for a thick or thin line of pigmentation at the level of the mucogingival junction. The pigmented zone is symmetric and the color uniform.

Category 4: Pigmentation is spread over the mucosa. It is asymmetric, patchy, and irregular. The color can be dark at one tooth and pink at the adjacent tooth.

Category 5: Mucosa is completely pink with the exception of a number of symmetric "islands" of pigmentation between anterior teeth. The patches are localized and dark, in contrast to the surrounding (pink) tissue. These patches do not extend to the gingiva. Category 6: Mucosa is completely pink and there are no signs of melanin pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients were free from any systemic disease as evidenced by Burkett's oral medicine health history questionnaire Greenberg et al.,2012.
* Patients with physiologic gingival hyperpigmentation in the aesthetic zone.

Exclusion Criteria:

* Smokers.
* Pregnant and lactating women.
* Drugs intake which associates with gingival melanin pigmentation such as Antimalarials drugs, phenothiazines and oral contraceptives.
* Pathologies that cause gingival pigmentation (e.g.: Addison's disease, Albright's syndrome, Kaposi sarcoma)
* Patients with periodontal disease.
* Physical or mental impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: population of any age except children that will seeking treatment at the dental clinics
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
pigmentation distribution | baseline
  to evaluate distribution of gingival pigmentation using Hedin melanin index and de Krom classification
  Hedin melanin index:
  Used for evaluation of the distribution of pigmentation in the gingiva. It is scored as 0= absence of gingival pigmentation.
  1. One or two isolated units of interdental papillae exhibit pigmentation.
  2. Three or more distinct units of interdental papillae exhibit pigmentation.
  3. continuous band of pigmented gingiva of short length. 4 = a broad band of continuous pigmented gingiva situated between the canines. de Krom classification: The de Krom classification has been invented to determine the distribution of pigmentation as follows:
     * Category 1: A wide band of pigmentation entirely encircles the dentition, exhibiting a distinct apical contour. The mucosa is pink above the mucogingival junction. The color of the gingiva may range from dark to light brown. The band is symmetrical, and its color is uniform.
     * Category 2: A narrow band of non-pigment
pigmentation intensity | baseline
  by using Dummet Oral Pigmentation Index (DOPI)
  This was used to evaluate the intensity of gingival pigmentation as follows:
  0= Absence of clinical pigmentation (pink-colored gingiva)
  1. Mild clinical pigmentation (light brown color)
  2. Moderate clinical pigmentation (medium brown or a combination of pink and brown color) 3 = Significant clinical pigmentation (dark brown or bluish-black color)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No